CLINICAL TRIAL: NCT01575639
Title: Randomized Trial of High Dose (4mg/kg) Versus Usual Dose (2mg/kg) Oral Prednisolone in the Treatment of Infantile Spasms.
Brief Title: Prednisolone in Infantile Spasms- High Dose Versus Usual Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Satinder Aneja, Director Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDIS
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Infantile Spasms; West Syndrome
MeSH Terms: conditions — Spasms, Infantile | interventions — Prednisolone

ARMS (2):
- High dose (Experimental): Oral Prednisolone will be given at dose of 4 mg/kg/day for 14 days
  Interventions: Drug: Oral prednisolone
- Usual dose (Active Comparator): Oral prednisolone will be given at dose of 2 mg/kg/day for 14 days
  Interventions: Drug: Oral prednisolone

INTERVENTIONS:
Drug: Oral prednisolone — Dose will be different in the two groups. the high dose group will receive 4 mg/kg/day. The usual dose group will receive 2 mg/kg/day

SUMMARY:
Infantile spasms comprise a difficult to treat type of epilepsy in young children. Hormonal treatment, i.e. Prednisolone and ACTH are considered the treatment of choice. There is no consensus on the dosage of Prednisolone required for the treatment of infantile spasms. Recent data has shown that a high dose (4 mg/kg/day) may be more efficacious than the usual dose (2 mg/kg/day). However, there are no randomized controlled trials comparing these doses. A higher steroid dose may also be associated with more side effects. Therefore, this study was planned to compare the efficacy and tolerability of the high dose versus the usual dose in children with infantile spasms, in a randomized open-label trial design

ELIGIBILITY:
Inclusion Criteria:

- Children aged 3 months to 2 years presenting with epileptic spasms (at least 1 cluster/day) with EEG evidence of hypsarrhythmia or its variants

Exclusion Criteria:

1. Children with active systemic illness
2. Children with evidence of active tuberculosis
3. Severe Acute Malnutrition ad defined by WHO (visible wasting/Mid Upper Arm Circumference < 11 cm/pedal edema/Weight for height < 3 SD)
4. Children with recurrent illness/chronic systemic illness

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children who achieved spasm freedom (for at least 48 hours) as per parental reports on day 14 . | 14 days

SECONDARY OUTCOMES:
Proportion of children with adverse effects | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Satinder Aneja, MD, Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College and Associated Kalawati Saran Children's Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Chellamuthu P, Sharma S, Jain P, Kaushik JS, Seth A, Aneja S. High dose (4 mg/kg/day) versus usual dose (2 mg/kg/day) oral prednisolone for treatment of infantile spasms: an open-label, randomized controlled trial. Epilepsy Res. 2014 Oct;108(8):1378-84. doi: 10.1016/j.eplepsyres.2014.06.019. Epub 2014 Jul 5. PMID 25048310